CLINICAL TRIAL: NCT04256772
Title: Anti-IL5 and Other Biotherapies in Cystic Fibrosis in French CF Centers : MAB-CF Cohort
Brief Title: Anti-IL5 and Other Biotherapies in Cystic Fibrosis
Acronym: MAB-CF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0563
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
Keywords: CYSTIC FIBROSIS; BIOTHERAPY; ANTI-IL5; BENRALIZUMAB; APBA; SEVERE ASTHMA
MeSH Terms: conditions — Cystic Fibrosis; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our project is to describe retrospectively and prospectively CF patients treated with biotherapy in French CF centers.

Main objective: To describe the clinical and paraclinical course of CF patients before and after treatment with anti-IL5 and other biotherapies since 2019.

Secondary objective: To describe adverse events potentially related to the biotherapies.

DETAILED DESCRIPTION:
•Background: ABPA and asthma associated with cystic fibrosis impact the CF course with a more rapid decline in lung function.

Corticosteroid therapy can be harmful and must be avoid in CF to prevent diabetes, osteoporomalacia or mycobacterium infections.

Monoclonal antibodies have the marketing authorization for severe uncontrolled asthma and, up to now, some CF patients with ABPA or severe asthma and high plasma IgE levels benefit from omalizumab.

Anti-Il5 agents are available since February 2019 and have demonstrated their efficacy in severe and hypereosinophilic asthma control (plasma eos.>300mmol/L).

Some patients with CF who have severe asthma or ABPA are still poorly controlled despite Omalizumab with other treatments (steroids and/or azoles). Some of them have persistent hypereosinophilia suggesting a possibility to treat with antiIL5 antibodies.

About 5% of patients have biotherapy treatment criteria, some have already received it, others are elective to such treatment and will receive in the future.

Methods:

Our project is to describe retrospectively and prospectively the clinical history of CF patients eligible for biotherapy in French CF centers.

Main objective: To describe the clinical and paraclinical course of CF patients before and after treatment with anti-IL5 and other biotherapies since 2019.

Secondary objective: To describe any adverse events potentially related to the biotherapies.

ELIGIBILITY:
Inclusion criteria:

* Cystic fibrosis (2 known variants)
* Age ≥ 6 years
* Plasma hypereosinophilia ≥ 300/µl
* Uncontrolled ABPA or uncontrolled asthma, or failure of other biotherapy (intolerance, ineffectiveness)

Exclusion criteria

- Refusal to participate in this research

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients (2 known variants) with hypereosinophilia ≥ 300/µl and uncontrolled ABPA or uncontrolled asthma, or failure of other biotherapy (intolerance, ineffectiveness)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution | 1 day
  Physical examination (height in centimeters, weight in kilograms, numerical scales in score, temperature in degrees, SaO2 in percentage).
  Defines the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis To assess the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis
Spirometry in liters or percentage evolution | 1 day
  Spirometry in liters or percentage Defines the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis
Biology evolution | 1 day
  Biology (leukocyte formula in 10^9/L, IgE tot, IgE spe, sputum microbiology) Defines the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis
concomitant therapy evolution | 1 day
  concomitant therapy Defines the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis
CFQR and SNOT22 evolution | 1 day
  CFQR and SNOT22 questionnaires in score Defines the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis
exacerbation evolution | 1 day
  Defines the effectiveness of anti-inflammatory biotherapy in patients with cystic fibrosis

SECONDARY OUTCOMES:
Number of any adverse event reported during biotherapy treatments | 1 day
  Describe any adverse event potentially related to biotherapies. description of any adverse event reported during biotherapy treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael CHIRON, PU-PH, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC